CLINICAL TRIAL: NCT05351190
Title: Community Glucose Monitoring (CGM) Project
Brief Title: Community Glucose Monitoring Project
Acronym: CMGProject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Blanchard Valley Health System (Other)
Responsible Party: Principal Investigator, Thomas Grace, MD, Principal Investigator, Blanchard Valley Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-2021-169
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Other): All participants will be given a rtCGM (Dexcom G6) to assess their glycemic control.
  Interventions: Device: Dexcom G6 CGM

INTERVENTIONS:
Device: Dexcom G6 CGM — rtCGM to be worn by user continuously for the duration of the 12 month study

SUMMARY:
The investigators believe that addition of real time continuous glucose monitoring (RT-CGM) improves glycemic outcome in patients with Type 2 diabetes compared to self-monitored blood glucose (SMBG), for patients who are not at target A1C regardless of treatment modality.

The investigators aims to assess glycemic and quality of life (QoL) benefits of adding and using RT-CGM patients with Type 2 Diabetes Mellitus (T2DM), not at their A1C goal and relying on SMBG for diabetes-management decisions.

DETAILED DESCRIPTION:
Prescreened and eligible subjects will obtain CGM and basic CGM education upon enrollment.

They will initially be given three months of CGM supplies and return to the study center every 3 months for more supplies. In addition, baseline data and labs will be collected at visits.

All subjects will return to the clinic after every three months for assessment and assignment of three more months of CGM supplies. This will repeat for a 12 month period.

Patient reported outcome (PRO) measurements will be obtained at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of T2DM
3. Followed regularly by a physician with at least 2 office visits in last year as documented by clinical history
4. Sub-optimal glycemic control, defined as persistent hyperglycemia, confirmed initially by historical or local (POC or site's lab) A1C of ≥7.7% NOTE: Use of a historical local A1C test must be within 1 month of study entry.
5. Desire to lower A1C such as a goal of 7%
6. Stable control of diabetes, as determined per investigator assessment
7. Willing to wear a CGM

Exclusion Criteria:

1. Use of personal RT-CGM 3 months prior to study entry (professional CGM use is allowed, whether it was blinded or un-blinded)
2. Current or anticipated acute uses of glucocorticoids (oral, injectable, or IV), that will affect glycemic control and impact A1C - such as frequent steroid bursts required for inflammatory arthritis or inflammatory bowel disease, recurrent lumbar epidural steroid injections, etc. (Long-term stable glucocorticoid doses are allowed, such as when used for the treatment of rheumatoid arthritis or Addison's disease).
3. Pregnancy (as demonstrated by a positive test at study entry screening) or are planning to become pregnant during the study
4. Medical conditions that, per investigator determination, make it inappropriate or unsafe to target an A1C of <7%, such as, but not limited to, recent cardio- or cerebro- vascular disease, malignancy, severe recurrent hypoglycemia, or cognitive decline
5. History of visual impairment which would hinder subject's participation in the study and perform all study procedures safely, as determined by investigator
6. History of psychiatric, psychological disorder, or psycho-social issues that could limit adherence to the required study tasks
7. Renal disease defined as estimated Glomerular Filtration Rate (eGFR) <45)
8. Extensive skin changes/disease that preclude wearing the sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis)
9. Known allergy to medical-grade adhesives
10. Current participation in another investigational study (must have completed any previous studies at least 30 days prior to being enrolled in this study)
11. Currently abusing illicit drugs, alcohol, or prescription drugs
12. Any condition per investigator assessment, that could impact reliability of the A1C measurement, such as (but not limited to) hemoglobinopathy, hemolytic anemia, chronic liver disease; chronic GI blood loss, recent red blood cell transfusion or erythropoietin administration within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
A1c | Baseline to 3 months
  Record Changes in HgbA1c
A1c | Baseline to 6 months
  Record Changes in HgbA1c
A1c | Baseline to 9 months
  Record Changes in HgbA1c
A1c | Baseline to 12 months
  Record Changes in HgbA1c

SECONDARY OUTCOMES:
Weight | Baseline to 3 months
  Record Changes
Weight | Baseline to 6 months
  Record Changes
Weight | Baseline to 9 months
  Record Changes
Weight | Baseline to 12 months
  Record Changes
BMI | Baseline to 3 months
  Record Changes
BMI | Baseline to 6 months
  Record Changes
BMI | Baseline to 9 months
  Record Changes
BMI | Baseline to 12 months
  Record Changes
Percent Time in Range (70-180 mg/dl) | Baseline to 3 months
  Record Changes
Percent Time in Range (70-180 mg/dl) | Baseline to 6 months
  Record Changes
Percent Time in Range (70-180 mg/dl) | Baseline to 9 months
  Record Changes
Percent Time in Range (70-180 mg/dl) | Baseline to 12 months
  Record Changes
Percent Time in Hypoglycemia (<70 mg/dl) | Baseline to 3 months
  Record Changes
Percent Time in Hypoglycemia (<70 mg/dl) | Baseline to 6 months
  Record Changes
Percent Time in Hypoglycemia (<70 mg/dl) | Baseline to 9 months
  Record Changes
Percent Time in Hypoglycemia (<70 mg/dl) | Baseline to 12 months
  Record Changes
Percent Time in Hyperglycemia (>180 mg/dl) | Baseline to 3 months
  Record Changes
Percent Time in Hyperglycemia (>180 mg/dl) | Baseline to 6 months
  Record Changes
Percent Time in Hyperglycemia (>180 mg/dl) | Baseline to 9 months
  Record Changes
Percent Time in Hyperglycemia (>180 mg/dl) | Baseline to 12 months
  Record Changes
Quality of Life - GMSS T2DM Version | Baseline to 6 months
  Record Changes in QoL
Quality of Life - GMSS T2DM Version | Baseline to 12 months
  Record Changes in QoL

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Grace, MD, Principal Investigator — Hancock County Health Department
Locations (1):
- Hancock County Health Department, Findlay, Ohio, United States

IPD SHARING:
Plan to Share IPD: No